CLINICAL TRIAL: NCT00243516
Title: Randomized, Controlled Trial for the Use of Pretest Probability to Reduce Unnecessary Testing for Low-Risk Patients With Chest Pain
Brief Title: Trial for the Use of Pretest Probability to Reduce Unnecessary Testing for Low-Risk Patients With Chest Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PREtest Consult (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2005-10-17; First posted 2005-10-24 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2006-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Emergency Department; Chest Pain Evaluation Unit; Overtesting; Chest Pain Protocol; Myocardial Infarction; Medical Malpractice
MeSH Terms: conditions — Acute Coronary Syndrome; Emergencies; Myocardial Infarction

INTERVENTIONS:
Device: PREtest Consult

SUMMARY:
The purpose of this study is to evaluate if the implementation of quantitative pretest probability assessment will significantly reduce the unnecessary use of the intra-emergency department chest pain center. Specifically, the study will examine whether the PREtest Consult acute coronary syndrome (ACS) pretest probability assessment system can significantly reduce the use of chest pain unit evaluation in very low risk emergency department (ED) patients, can safely discharge patients with a pretest probability ≤ 2.0%, can reduce unnecessary procedures and lower hospital costs and will examine patient satisfaction of patients with whom pretest probability assessment was used compared to those with whom it was not used.

The researchers hypothesize that patients in the control group of the study will have statistically significant reductions in mean time spent in the emergency department, mean charges billed to the patient or their insurance carrier, hospital length of stay, mean number of procedures or tests performed without a statistically significant change in patient satisfaction or adverse outcome.

DETAILED DESCRIPTION:
Chest pain represents the second most frequent complaint among the 110 million persons who visit emergency departments in the U.S. each year. Perceived medicolegal risk compels emergency physicians to overtest for possible acute coronary syndrome (ACS), contributing to more than $20 billion in unnecessary diagnostic testing each year. The hypothesis of the present work states that quantitative pretest probability assessment can significantly and safely increase the proportion of very low risk patients with symptoms of ACS who are discharged from one emergency department. Quantitative pretest probability will be assessed with the validated, commercially available PREtest Consult ACS software device, which employs computer assisted, attribute matching. This method matches an 8-component clinical profile from any individual patient to the same profile shared by patients who were previously evaluated for ACS and whose profiles are stored in a 14,800 patient reference database. Pretest probability estimates ≤ 2% will be considered "test negative." A phase II multicenter study found that when the ACS PREtest Consult produced a pretest probability of ACS ≤ 2.0% that the actual outcome of ACS at 45 days was 0.3% (95% CI 0 to 1.8%) compared with 0.4% (0 to 0.9%) for patients discharged after negative testing in a chest pain unit (CPU) that included serial biomarkers, overnight monitoring, and cardiologist-interpreted provocative testing. Over one-quarter of all patients referred to the CPU had an estimate ≤ 2%. The present study will randomize 400 ED patients with a non-diagnostic or normal ECG and a troponin test ordered into two groups:

1. a "show me", or disclosure group, in which patients and their clinicians will receive the output of the device, and
2. a "no show" or concealed group will receive no output.

The sample size will detect an 11.5% difference in rate of discharge between groups with α = 0.05 and β = 0.20. All discharged patients will undergo structured telephone and medical record follow-up at 7 and 45 days using validated methodology.

Primary outcome measures will evaluate the development of acute coronary syndrome.

Secondary variables will include:

1. Frequency of ACS, determined by blinded adjudicated review of follow-up data,
2. Rate of return to any ED for similar symptoms,
3. Patient satisfaction,
4. Charges.

Project significance includes the potential to reduce patient exposure to unnecessary invasive procedures and to save Medicare and other insurers over $100 million in unnecessary diagnostic testing each year in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patients aged > 17 who report a history of torso or arm discomfort within the past 24 hours.
* Physician orders an electrocardiogram and serum troponin measurement.
* Physician has undergone a 10 minute explanation session and has provided consent

Exclusion Criteria:

* 12-lead electrocardiogram (ECG) with ST deviation or T-wave changes that are interpreted by clinician as indicative of acute infarction or ischemia
* "Code STEMI" patients (patients with suspected acute myocardial infarction).
* Other primary diagnosis mandating admission (e.g., pneumonia, diabetic ketoacidosis, trauma)
* Patients with myocardial infarction, intracoronary stent placement, or coronary artery bypass grafting within the previous 30 days.
* Evidence of circulatory shock (SBP [systolic blood pressure] < 100 mmHg with symptoms defined by Jones)
* Cocaine use within the past 72 hours.
* A moderate to high-risk composite clinical picture that causes an emergency medicine specialist to consult a cardiologist.
* Homelessness, out-of-town residence or other condition known to preclude follow-up.
* Prisoners and pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-10; Study Completion 2007-10

PRIMARY OUTCOMES:
Documented myocardial infarction (ESC criteria)
Death thought to be from ACS (autopsy not required)
Need for revascularization (stent or surgical) within 45 days
Cardiac catheterization demonstrating

SECONDARY OUTCOMES:
Percentage of patients deemed very low risk (pretest probability less than 2%) by the physician or the PREtest Consult ACS platform during the index visit
Percentage of patients discharged without admission to the hospital or emergency department chest pain unit during the index visit
Length of stay for the index visit to the emergency department
Incidence of stress testing, cardiac imaging and cardiac catheterization during the index visit and in the 45 days following the index visit
Hospital charges billed to each patient or their insurance provider for the index visit
Rate of reimbursement to the hospital for the index visit of each patient
Patient satisfaction as recorded by a survey instrument during a phone interview seven (7) days post-index visit

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Kline, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States